CLINICAL TRIAL: NCT01894490
Title: Randomized Clinical Trial: Nasoenteric Catheter or Jejunostomy as a Route For Nutrition After Major Upper Gastrointestinal Operations
Brief Title: Randomized Clinical Trial: Nasoenteric Catheter or Jejunostomy
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, MD, PhD, Federal University of Minas Gerais
Other Study IDs: 301/08
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Complications After Gastrointestinal Operations
Keywords: Gastrointestinal surgery, complications, length of hospital stay, mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Jejunostomy: Patients who received a jejunostomy
- Nasojejunal catheter: Patients who received a nasojejunal catheter

SUMMARY:
Curative treatment of upper gastrointestinal tract neoplasms is complex and associated with high morbidity and mortality. In general, the patients are already malnourished, and early postoperative enteral nutrition is recommended. However, there is no consensus concerning the best enteral access route in these cases.

DETAILED DESCRIPTION:
A prospective randomized trial with patients undergoing esophagectomy, total gastrectomy or pancreaticoduodenectomy to asses the outcomes of either jejunostomy placement or catheter placement

ELIGIBILITY:
Inclusion Criteria:

* age over 18,
* gastrointestinal resections

Exclusion Criteria:

* age under 18,
* no gastrointestinal procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal disorders undergoing major abdominal operations
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Complications | 30 day
  Follow up patients after undergoing operation up to 30 days

SECONDARY OUTCOMES:
Length of hospital stay | 30 days
  Length of hospital stay in both groups

OTHER OUTCOMES:
Mortality | 30 day
  Mortality due to surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Maria Isabel TD Correia, MD, PhD, Study Director — Federal University of Minas Gerais
Locations (1):
- Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil